CLINICAL TRIAL: NCT07208981
Title: A Prospective Multicenter Study of Orelabrutinib Combined With Zebetuzumab and Lenalidomide or Bendamustine Combined With Rituximab for the Treatment of Newly Diagnosed MZL
Brief Title: Orelabrutinib Combined With Zebetuzumab and Lenalidomide for the Treatment of Newly Diagnosed MZL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Optional
Record Dates: First submitted 2025-09-18; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-08

CONDITIONS: Marginal Zone Lymphoma(MZL)
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — orelabrutinib; Lenalidomide; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of orelabrutinib combined with zebetuzumab and lenalidomide (Experimental)
  Interventions: Drug: Orelabrutinib; Drug: Zebetuzumab; Drug: Lenalidomide
- Group of bendamustine combined with rituximab (Active Comparator)
  Interventions: Drug: Bendamustine + Rituximab

INTERVENTIONS:
Drug: Orelabrutinib — Induction treatment phase (a total of 6 cycles, each cycle lasting 28 days), Orelabrutinib (150 mg, d1-d28). Maintenance phase (a total of 24 cycles, each cycle lasting 28 days), Orelabrutinib (150 mg, d1-d28). Patients who achieve complete remission (CR) or partial remission (PR) after 6 cycles will decide whether to undergo maintenance therapy based on the investigator's choice.
  Arms: Group of orelabrutinib combined with zebetuzumab and lenalidomide
Drug: Zebetuzumab — Induction treatment phase (a total of 6 cycles, each cycle lasting 28 days), Zebetuzumab (375 mg/m2, d1/C1-C6).
  Arms: Group of orelabrutinib combined with zebetuzumab and lenalidomide
Drug: Lenalidomide — Induction treatment phase (a total of 6 cycles, each cycle lasting 28 days), Lenalidomide (20 mg, d1-d21).
  Arms: Group of orelabrutinib combined with zebetuzumab and lenalidomide
Drug: Bendamustine + Rituximab — Treatment period (a total of 6 cycles, each cycle lasting 28 days), Bendamustine (90 mg/m2, d1-2), Rituximab (375 mg/m2, d1/C1-6).
  Arms: Group of bendamustine combined with rituximab

SUMMARY:
This is an open-label, multicenter, phase 2, non-randomized study aiming to evaluate the efficacy and safety of orelabrutinib combined with zebetuzumab and lenalidomide or bendamustine combined with rituximab in the treatment of newly diagnosed marginal zone lymphoma (MZL).

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-75 years, gender not restricted;
* 2. Histopathologically confirmed CD20-positive marginal zone lymphoma includes MALT, SMZL, and NMZL; at least one measurable lesion;
* 3. Indication for treatment

  * 3.1. Initial diagnosis II 2 or IIE or IV stage gastric MALT treatment indications. Including: ① Meeting the inclusion criteria for clinical trials; ② Presence of lymphoma-related clinical symptoms; ③ Gastrointestinal bleeding (bleeding condition controlled or assessed by the investigator for suitability of inclusion); ④ End-organ damage; ⑤ Large mass; ⑥ Persistent or rapid disease progression; ⑦ Patient's willingness;
  * 3.2. Recommendations for treatment indications of newly diagnosed stage III-IV non-gastric MALT and NMZL. The GELF criteria, similar to those used for follicular lymphoma, include: ① The presence of ≥3 distinct regions of involved lymph nodes, with each involved lymph node having a diameter of ≥3 cm; ② The presence of any lymph node or extranodal lesion with a diameter >7 cm; ③ The presence of B symptoms; ④ Splenomegaly; ⑤ Symptoms of organ compression, pleural or peritoneal effusion; ⑥ Cytopenia caused by the disease; ⑦ Persistent or rapid disease progression, with tumor size increasing by 20%-30% within 2-3 months or approximately 50% within 6 months; ⑧ Meeting the inclusion criteria for clinical trials;
  * 3.3. Recommended indications for the treatment of newly diagnosed SMZL. Including: ① Progressive or painful splenomegaly; ② Symptomatic or progressive cytopenia such as HB<100g/L, PLT<80×10^9/L, absolute neutrophil count (ANC)<1.0×10^9/L (note to differentiate from cytopenia caused by autoimmune factors);
* 4. Without prior systemic treatment, may include MZL (marginal zone lymphoma) that has progressed, relapsed, or is unsuitable for local treatment after previous local therapy (local treatment includes surgery, radiotherapy, anti-Helicobacter pylori therapy for at least 12 months, or anti-hepatitis C therapy);
* 5. ECOG performance status score 0-2 points
* 6. The main organ functions meet the following criteria (except for SMZL, which is judged separately by the investigator to meet treatment requirements): Complete blood count: Absolute neutrophil count ≥1.5×10^9/L, platelets ≥75×10^9/L, hemoglobin ≥75g/L; if accompanied by bone marrow involvement, absolute neutrophil count ≥1.0×10^9/L, platelets ≥50×10^9/L, hemoglobin ≥50g/L; Blood biochemistry: Total bilirubin ≤ 1.5 times ULN, AST or ALT ≤ 2 times ULN; serum creatinine ≤ 1.5 times ULN; serum amylase ≤ ULN; creatinine clearance rate ≥ 60 mL/min;
* 7. Coagulation function: International Normalized Ratio (INR) ≤1.5 times ULN;
* 8. Expected survival time ≥ 12 months;
* 9. Voluntarily sign a written informed consent before trial screening.

Exclusion Criteria:

* 1. Currently or previously diagnosed with other malignancies, unless radical treatment has been performed and there is evidence of no recurrence or metastasis within the past 5 years, excluding cured cervical carcinoma in situ, basal cell carcinoma of the skin, and localized squamous cell carcinoma of the skin;
* 2. Lymphoma involving the central nervous system or transforming to a higher grade;
* 3. Uncontrolled or significant cardiovascular diseases, including: a) Occurrence of New York Heart Association (NYHA) Class III-IV congestive heart failure, unstable angina, myocardial infarction within 6 months prior to the first administration of the investigational drug, or the presence of treatable arrhythmias at screening, with left ventricular ejection fraction (LVEF) <50%; b) Primary cardiomyopathies (such as dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, unclassified cardiomyopathy); c) A clinically significant history of QTc interval prolongation, or QTc interval during the screening period >470ms for females and >450ms for males; d) Subjects with symptomatic or medication-requiring coronary heart disease; e) Suffering from uncontrolled hypertension (blood pressure remains uncontrolled after more than one month of using a reasonable and tolerable dosage of three or more antihypertensive drugs (including diuretics) based on lifestyle improvements, or blood pressure can only be effectively controlled by taking four or more antihypertensive drugs);
* 4. Active bleeding within 2 months prior to screening, or currently taking anticoagulants, or deemed by the investigator to have a clear bleeding tendency;
* 5. History of deep vein thrombosis or pulmonary embolism in the past six months;
* 6. Underwent major surgery within 6 weeks prior to screening or minor surgery within 2 weeks prior to screening. Major surgery refers to procedures performed under general anesthesia, but endoscopic examinations for diagnostic purposes are not considered major surgery. The insertion of vascular access devices is exempt from this exclusion criterion;
* 7. Active infection or uncontrolled HBV (HBsAg positive and/or HBcAb positive with HBV DNA titer positive), HCV RNA positive, HIV/AIDS, or other severe infectious diseases;
* 8. Currently, there are subjects with severe pulmonary function impairment due to conditions such as pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, and drug-related pneumonia: FEV1% or DLCO (or DLCO/VA) %pred < 40% (with severe pulmonary ventilation and gas exchange dysfunction);
* 9. Pregnant, lactating women and childbearing age subjects unwilling to use contraception;
* 10. Need to continuously take medications with moderate to strong inhibitory or strong inducing effects on cytochrome P450 CYP3A;
* 11. The investigator considers other conditions unsuitable for participating in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2031-06-01 (Estimated)

PRIMARY OUTCOMES:
3-year PFS rate | From the first dose of treatment to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 66 months.
  PFS is defined as the first dose of treatment to the date of first documented progression or date of death from any cause, whichever occurs first. 3-year PFS rate will be estimated by Kaplan-Meier.

SECONDARY OUTCOMES:
Overall response rate (ORR) | On Day 1 of Cycle 4, Day 1 of Cycle 7, Day 1 of Cycle 13, Day 1 of Cycle 19, Day 1 of Cycle 25, Day 1 of Cycle 31 (each cycle is 28 days).
  Overall response rate is the proportion of patients who achieve either a complete or partial response to treatment defined by the Lugano classification criteria for lymphoma response evaluation (2014 edition)/GELA (gastric MALT).
Rate of best overall response (BOR) | On Day 1 of Cycle 4, Day 1 of Cycle 7, Day 1 of Cycle 13, Day 1 of Cycle 19, Day 1 of Cycle 25, Day 1 of Cycle 31 (each cycle is 28 days).
  The rate of best overall response is the proportion of patients who achieve their best recorded response (complete or partial) to treatment at any time during the study.
Time to response (TTR) | On Day 1 of Cycle 4, Day 1 of Cycle 7, Day 1 of Cycle 13, Day 1 of Cycle 19, Day 1 of Cycle 25, Day 1 of Cycle 31 (each cycle is 28 days).
  Time to response is the duration from the start of treatment to the first documentation of a complete or partial response.
Progression-free survival (PFS) rate | From the first dose of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 66 months.
  PFS is defined as the time from the first dose of treatment until the date of first documented progression or date of death from any cause, whichever occurs first. For subjects without progression, relapse, or death at the time of analysis, EFS will be censored at the last assessment date.
Overall survival (OS) rate | From the first dose of treatment until the date of death from any cause, assessed up to 66 months.
  OS is defined as the time from the first dose of treatment until the date of death from any cause, assessed up to 66 months. Subjects who remain alive at the time of analysis will be censored at the last known alive date of the subject.
Rate of progression of disease within 24 months (POD24) | On Day 1 of Cycle 4, Day 1 of Cycle 7, Day 1 of Cycle 13, Day 1 of Cycle 19, Day 1 of Cycle 25, Day 1 of Cycle 31 (each cycle is 28 days).
  Progression of disease within 24 months is defined as patients whose disease relapse or progress within 24 months of first treatment.
Quality of life (FACT-Lym) | On Screening, Day 1 of Cycle 1, Day 1 of Cycle 4, Day 1 of Cycle 7, Day 1 of Cycle 13, Day 1 of Cycle 19, Day 1 of Cycle 25, Day 1 of Cycle 31 (each cycle is 28 days).
  FACT-Lym (Functional Assessment of Cancer Therapy-Lymphoma) is a validated questionnaire that measures health-related quality of life in patients with lymphoma, covering physical, social/family, emotional, and functional well-being, along with lymphoma-specific symptoms and concerns. FACT-Lym has 42 items, and scores of every item range from 0 to 4, with higher scores indicating better quality of life.
Adverse Events | From screening to 3 years after the end of maintenance therapy.
  All treatment-emergent AEs will be included in the analysis. For each AE, the number and percentage of subjects who experience at least one occurrence of the given event will be summarized. The number and percent of subjects with TEAEs will be summarized according to intensity (CTCAE, v5) for hematologic toxicity, and drug relationship, as well as categorized by system organ class and preferred term. Summaries, listings, datasets, or subject narratives may be provided, as appropriate, for those subjects who die, who discontinue treatment due to an AE, or who experience a severe AE or a SAE.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Jiangsu Province Hospital, Nanjing, Jiangsu, China